CLINICAL TRIAL: NCT05399342
Title: Left Atrial Appendage Occlusion III Extended Follow Up
Brief Title: Left Atrial Appendage Occlusion Study III Extended Follow Up
Acronym: LAAOSIIIX
Status: Withdrawn | Type: Observational
Why Stopped: Did not receive grant funding to conduct the study
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: LAAOSIII Extension
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Left Atrial Appendage Occlusion
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAAOS III Extended Follow-Up Cohort: Patients randomized into the LAAOS III trial who have consented to longer term observational follow-up. There is no intervention in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Patients in the LAAOS III trial either had or did not have their left atrial appendage occluded at the time of surgery in that trial. No further intervention is required in this cohort, it is observational follow-up only.

SUMMARY:
LAAOS III Extension is a longer term follow-up of an international cohort study of patients who were enrolled in the Left Atrial Appendage Occlusion Study (LAAOS III) trial.

DETAILED DESCRIPTION:
The association between atrial fibrillation and heart failure has been well established. Although the causal relationship between the two clinical entities has not been fully elucidated, atrial fibrillation is believed to cause heart failure via several mechanisms: 1) increased heart rate resulting in shorter diastolic filling time and lower cardiac output; 2) reduced atrial contraction contribution to left ventricular filling, lowering cardiac output; and 3) tachycardia-induced cardiomyopathy from myocardial ischemia, myocardial energy depletion, and abnormal calcium regulation leading to left ventricular dilatation and reduced ejection fraction. These processes occur over time. It is also established that the left atrial appendage is a source of atrial natriuretic peptide, and it has been hypothesized that removal of the appendage might impair renal clearance of salt and water, increasing the risk of heart failure. A recent non-randomized study has supported this hypothesis. In LAAOS III, we did not observe an increase in hospitalization for heart failure, either early after surgery or during the 3.8 years of follow-up. However, an adverse impact on heart failure may appear over a longer follow-up period. We need to ensure we examine this patient population for the long-term impact of left atrial appendage occlusion on heart failure hospitalization to ensure we fully appreciate the benefit-risk balance of this intervention.

The extended follow-up of the LAAOS III trial aims to assess whether, in patients with a history of atrial fibrillation undergoing cardiac surgery for another indication, concomitant left atrial appendage occlusion decreases the risk of death and stroke on top of usual care including anticoagulation without increasing re-hospitalization for heart failure at a mean follow-up of 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant was enrolled in the LAAOS III trial
* Participant has provided written informed consent

Exclusion Criteria:

* Participant did not undergo the index LAAOS III cardiac surgery
* Participant underwent heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of participants of the Left Atrial Appendage Occlusion III trial (ClinicalTrials.gov ID: NCT01561651)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Mean follow up of 8 years after LAAOS III cardiac surgery
  The primary objective is to determine the impact of left atrial appendage (LAA) occlusion on all-cause mortality

SECONDARY OUTCOMES:
Impact of LAA occlusion on the incidence of ischemic stroke or or non-cerebral systemic embolism | Mean follow up of 8 years after LAAOS III cardiac surgery
  To examine the impact of LAA occlusion on the incidence of ischemic stroke or non-cerebral systemic embolism
Impact of LAA occlusion on re-hospitalization for heart failure | Mean follow up of 8 years after LAAOS III cardiac surgery
  Impact of LAA occlusion on re-hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, Principal Investigator — Population Health Research Institute; Emilie Belley-Côté, Principal Investigator — Population Health Research Institute